CLINICAL TRIAL: NCT07397572
Title: Prophylactic Oral Iron Supplementation for the Prevention of Iron Deficiency Anemia After Sleeve Gastrectomy: A Prospective Comparative Cohort Study
Brief Title: Iron Supplementation and Anemia After Sleeve Gastrectomy
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Eid Ali Ahmed Aziz, Lecturer, Cairo University
Other Study IDs: MS-679-2025
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Iron Deficiency Anemia; Obesity; Sleeve Gastrectomy
Keywords: Laparoscopic Sleeve Gastrectomy; Bariatric Surgery; Iron Deficiency Anemia; Iron Supplementation; Multivitamin; Morbid Obesity; Observational Study
MeSH Terms: conditions — Anemia, Iron-Deficiency; Obesity; Obesity, Morbid | interventions — Geritol; Minerals

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prophylactic Oral Iron Group: Patients from the bariatric surgery unit whose standard postoperative care includes a prophylactic oral iron regimen. This consists of Ferrodep® (30 mg elemental iron per capsule), one capsule every 12 hours (total 60 mg/day), in addition to a daily standard multivitamin.
  Interventions: Drug: Elemental Iron; Dietary Supplement: Multivitamin with Minerals
- Standard Multivitamin Group: Patients from the bariatric surgery unit whose standard postoperative care includes a daily standard multivitamin only (e.g., Centrum Silver®), which contains approximately 10 mg of iron. No additional prophylactic iron is routinely prescribed.
  Interventions: Dietary Supplement: Multivitamin with Minerals

INTERVENTIONS:
Drug: Elemental Iron — Prophylactic oral iron supplement (Ferrodep®), prescribed as part of the standard post-operative care protocol at the participating unit. Each capsule contains 30 mg of elemental iron. The regimen is one capsule every 12 hours, for a total daily dose of 60 mg elemental iron, taken in addition to a daily multivitamin.
  Groups: Prophylactic Oral Iron Group
Dietary Supplement: Multivitamin with Minerals — A standard daily multivitamin with minerals (Centrum Silver®), prescribed as part of the routine post-operative care. This formulation contains approximately 10 mg of elemental iron. For participants in this unit's protocol, no additional prophylactic iron is routinely prescribed.

SUMMARY:
The goal of this observational study is to learn if taking extra iron pills after weight loss surgery helps prevent low iron and anemia compared to just taking a standard multivitamin. The main question it aims to answer is:

Does a specific iron supplementation plan lower the number of patients who develop iron deficiency anemia in the 6 months after sleeve gastrectomy surgery?

Researchers will compare two groups of patients from different hospital units to see if the extra iron works:

Patients from one unit who take a prophylactic iron supplement (Ferrodep, 60 mg per day) in addition to their standard multivitamin.

Patients from another unit who take only a standard multivitamin (Centrum Silver).

Participants in this study will:

* Have their blood tested for iron and anemia levels before surgery, and again at 3 and 6 months after surgery, as part of their regular post-operative care.
* Be asked about their health and quality of life during follow-up clinic visits.
* Have their medical information from their hospital records reviewed by the study team to track their progress.

DETAILED DESCRIPTION:
Background and Rationale Iron deficiency anemia (IDA) is a prevalent and clinically significant long-term complication following Laparoscopic Sleeve Gastrectomy (LSG), the most commonly performed bariatric procedure worldwide. Despite universal multivitamin supplementation, the incidence of IDA rises steadily post-operatively, impacting patient quality of life, cognitive function, and healthcare utilization. A critical evidence gap exists regarding the efficacy of routine prophylactic oral iron supplementation compared to a strategy of standard multivitamin use with iron monitoring. Current guidelines lack consensus due to insufficient comparative long-term data. This study aims to provide high-level evidence to inform postoperative protocols by directly comparing these two distinct management strategies.

Study Design and Setting This is a prospective, observational, comparative cohort study conducted within the bariatric surgery units of Kasr Al-Ainy Hospital, Cairo University. The study leverages existing, routine clinical practices at two participating units, allowing for a real-world comparison of outcomes. Participants will be managed according to the standard post-operative supplementation protocol of their treating surgical unit; the research protocol does not assign interventions.

Study Cohorts

Eligible participants will be enrolled into one of two cohorts based on the standard care protocol of their surgical unit:

Prophylactic Iron Cohort: Patients whose standard care includes a daily prophylactic dose of 60 mg elemental iron (administered as Ferrodep®, 30 mg capsule every 12 hours) in addition to a daily standard multivitamin.

Standard Multivitamin Cohort: Patients whose standard care includes a daily standard multivitamin only (e.g., Centrum Silver®), which contains approximately 10 mg of iron, with no additional prophylactic iron.

Study Procedures and Assessments Consecutively enrolled patients scheduled for primary LSG will be assessed pre-operatively (baseline) and at 3 and 6 months post-operatively. Data collection will include standardized laboratory panels (hemoglobin, ferritin, iron studies, complete blood count indices), documentation of supplementation adherence, and patient-reported outcome measures. All primary and secondary outcome measures are pre-specified and listed in the designated module.

Statistical Considerations The primary outcome is the cumulative incidence of IDA at 6 months post-surgery, with IDA defined per protocol-specific laboratory criteria. Secondary outcomes include longitudinal changes in hematological parameters, adherence rates, and patient-reported fatigue. A sample size of 66 participants (33 per cohort) was calculated to provide 85% power to detect a significant difference in the primary outcome. Data will be analyzed using SPSS software with appropriate statistical tests for between-group comparisons, as detailed in the statistical analysis plan.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years scheduled to undergo primary laparoscopic sleeve gastrectomy (LSG).
* Capable of understanding and providing written informed consent for participation.
* Able and willing to commit to the 6-month post-operative follow-up schedule at the bariatric clinic.

Exclusion Criteria:

* Prior history of major gastrointestinal surgery (e.g., bowel resection, gastrectomy) that could independently affect iron absorption.
* Pre-existing malabsorptive conditions (e.g., inflammatory bowel disease, celiac disease).
* Diagnosis of other known forms of anemia (e.g., thalassemia, vitamin B12/folate deficiency, anemia of chronic disease) that would confound the diagnosis of iron deficiency anemia (IDA).
* Any condition that, in the investigator's judgment, would interfere with full participation in the study or pose a significant risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with morbid obesity scheduled to undergo primary laparoscopic sleeve gastrectomy (LSG) at the participating bariatric surgery units.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2026-01-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Iron Deficiency Anemia (IDA) at 6 Months | 6 Months Post-Surgery
  Proportion of participants diagnosed with IDA. Diagnosis requires: 1) Anemia (Hemoglobin <13 g/dL in males or <12 g/dL in females), AND 2) Iron Deficiency, defined by at least one of: serum ferritin <30 ng/mL, TIBC >450 µg/dL, or serum iron <75 µg/dL (male)/<60 µg/dL (female).

SECONDARY OUTCOMES:
Change in Hemoglobin Concentration | Baseline, 3 Months, 6 Months
  Mean change in hemoglobin concentration (g/dL) from baseline to follow-up.
Change in Serum Ferritin Level | Baseline, 3 Months, 6 Months
  Mean change in serum ferritin concentration (ng/mL) from baseline to follow-up.
Change in Transferrin Saturation (TSAT) | Baseline, 3 Months, 6 Months
  Mean change in Transferrin Saturation percentage, calculated from serum iron and TIBC.
Incidence of Isolated Iron Deficiency without anemia | 3 Months, 6 Months
  Proportion of participants with serum ferritin <30 ng/mL and normal hemoglobin (≥12 g/dL female, ≥13 g/dL male).
Rate of Oral Iron Intolerance | 6 Months Post-Surgery
  Proportion experiencing gastrointestinal effects leading to dose reduction, interruption, or discontinuation of iron.
Adherence to Oral Supplementation | 3 Months, 6 Months
  Adherence expressed as the percentage of prescribed doses taken, calculated from pill count at follow-up clinic visits.
Fatigue Severity Score] | Baseline, 3 Months, 6 Months
  Mean score on the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) scale.The FACIT-Fatigue scale consists of 13 items, with total scores ranging from 0 to 52, where higher scores indicate less fatigue and better quality of life.
Need for Therapeutic Iron Supplementation | 6 Months Post-Surgery
  Proportion of participants who require initiation of new therapeutic iron during follow-up per clinician judgment.

CONTACTS AND LOCATIONS:
Overall Officials: Aziz, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine Cairo University, Cairo, Al-Manial Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No